CLINICAL TRIAL: NCT02822781
Title: Chronic Rhinosinusitis Classification Proposal: Evaluation of the Severity and the Effectiveness of Medical and Surgical Treatments
Brief Title: Chronic Rhinosinusitis Classification Proposal
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: CLASSIFICATION RSC
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: RHINOPLASTY; NASAL SURGICAL PROCEDURES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — There is no intervention. The patients will receive common questionnaire usually used by doctors (SNOT 22). Some Data to describe the population are collected then.

SUMMARY:
Chronic rhinosinusitis (CRS) is a debilitating disease that remains (smell, nasal patency, flow) because currently treatment protocols available to us are with a limited efficacy. The assessment of the response to surgical treatment protocols and monitoring the become of patients treated with only drugs should allow investigators to identify the predictive patient's profile for the response. With this prospective data, this study would allow investigators to make a classification of Chronic rhinosinusitis.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is a debilitating disease that remains (smell, nasal patency, flow) because currently treatment protocols available to us are with a limited efficacy.

For many years, practitioners have tried to identify a universal therapeutic protocol. It turns out that no treatment (functional endoscopic surgery, antifungal therapy, medical treatment with antibiotics / corticosteroids) does not resolve all of the symptoms and their effectiveness is variable from one patient to another.

The most plausible explanation is that the term "rhinosinusitis" includes various different pathophysiological mechanism entities, requiring different treatment. Like certain skin or lung diseases, chronic inflammation of the sinuses may have different origins, allergic or extrinsic (infectious). It is therefore important to determine the type of inflammation responsible for adapting the management.

First, it is important to determine from all forms of CRS (with or without polyps), those associated with allergic inflammation and infectious ones. The presence or absence of polyps does not appear to be a determining factor of the type of inflammation. However, the criteria - allergy and asthma - could provide guidance to an allergic mechanism.

The study aims to distinguish different phenotypes CRS according to clinical, anatomical criteria and biological criteria. Clinical classification obtained would assess and predict more finely treatment response and target according to the phenotype, the best supported. Surgery is one of the therapeutic options in the treatment of rhinosinusitis, but the term satisfaction of healing and patient comfort is variable, a finer and precise distribution of patients will allow us to better predict the success of the surgery and therefore the offer targeted patients.

Primary objective :

To assess the response to surgical treatment of rhinosinusitis and the outcome of these patients in order to highlight predictors of success of surgery.

Secondary objectives:

Assess chronic rhinosinusitis phenotype by score SNOT 22 (importance of symptoms) which assesses the average severity of different groups Assessing the future of non-operated patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral chronic rhinosinusitis evolving for more than 3 months with diffuse sinus opacities scanner.

Exclusion Criteria:

* Rhino Sinusitis unilateral
* Background total or functional ethmoidectomy (but not polypectomy)
* immunodeficiency or immunosuppression in patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bilateral chronic rhinosinusitis evolving for more than 3 months with diffuse sinus opacities scanner.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Assessment of change of the SNOT 22 score with a significant improvement from a minimal decrease of 10 points | Day1, Month 6
  Assessment of change of the SNOT 22 score with a significant improvement from a minimal decrease of 10 points

SECONDARY OUTCOMES:
Assessment of change of endoscopic nasal in consultation | Day1, Month 6

CONTACTS AND LOCATIONS:
Overall Officials: SAUVAGET Elisabeth, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (3):
- France (3):
  - Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region
  - L'Institut Arthur vernes, Paris, Île-de-France Region
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided